CLINICAL TRIAL: NCT06278012
Title: Development, Validity and Reliability of Atılım Kinesiophobia Scale
Brief Title: Development of Atılım Kinesiophobia Scale
Status: Recruiting | Type: Observational
Sponsor: Atılım University (Other)
Responsible Party: Principal Investigator, NAİME ULUG, Assistant Professor, Atılım University
Other Study IDs: E-59394181-604.01.02-32288
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-02

CONDITIONS: Kinesiophobia; Acute Pain; Chronic Pain; Fear of Movement
Keywords: pain, fear of movement, kinesiophobia, Turkish scale
MeSH Terms: conditions — Kinesiophobia; Acute Pain; Chronic Pain; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

Kinesiophobia or fear of movement, is defined as an excessive and irrational fear of physical movement to avoid painful injury, harm or re-injury. The existing scales measuring kinesiophobia are thought to have some limitations (the difficulty of patients to understand and answer the questions, the presence of questions that are not suitable for the patient's condition). These questionnaires may not have specific questions enough to assess fear of movement in different patient populations.

Aim: The aim of this study is to develop and validate the Turkish Atılım Kinesiophobia Scale.

Material/method:

In the first stage of the study, research on kinesiophobia was reviewed and a total of 38 questions were created for the scale. The questions were submitted to the opinion of 11 experts working in the physiotherapy and rehabilitation field. Then A total of 100 patients with acute and chronic musculoskeletal pain completed the Turkish Atılım Kinesiophobia Scale and Tampa Scale of Kinesiophobia.

DETAILED DESCRIPTION:
Kinesiophobia, or fear of movement, is defined as an excessive and irrational fear of physical movement to avoid painful injury, harm or re-injury. The prevalence of kinesiophobia in chronic painful conditions, especially musculoskeletal pain, has been reported to be between 50% and 70%. Pain-induced fear of movement or kinesiophobia negatively affects response to treatment, recovery and mobility in patients with injury, acute-chronic pain and in patients undergoing rehabilitation. Early and accurate detection of the presence of pain-induced fear of movement and education about kinesiophobia will be beneficial in the rehabilitation and recovery processes of patients (treatment processes will be shortened and recovery success will increase). Today, existing scales measuring kinesiophobia are thought to have some limitations. Especially the Tampa Kinesiophobia Scale is one of the most frequently used scales in the literature to assess kinesiophobia. This scale, whose Turkish validity and reliability study was conducted by the project coordinator and his colleagues, is used by many health professionals working in this field, especially physiotherapists in our country. However, in the studies in the literature and in the previous research of the project coordinator, it was determined that there were limitations and deficiencies related to the scale (the difficulty of patients to understand and answer the questions, the presence of questions that are not suitable for the patient's condition, the lack of questions for patient groups with different characteristics, etc.).

For these reasons, it was thought that there was a need to develop a new scale using a simple language that patients could easily understand. The new scale planned to be developed is intended to be able to measure kinesiophobia by including questions for patients with acute, chronic pain, post-surgical pain, neurological and geriatric patients who receive services in the field of physiotherapy and rehabilitation in the clinic. In addition, the scale to be designed is planned to evaluate the patients' fear of movement with biological, psychological and social reasons according to the International Classification of Functioning, Disability and Health (ICF) model.

Method:

This research is planned as a validity and reliability study in which the Turkish Atılım Kinesiophobia Scale will be developed. After the literature review on the subject, a pool of questions appropriate to the content of the ICF, which evaluates kinesiophobia with patient statements taken from the literature, will be created. Considering the differences in the disease status of the patients, questions for different patient groups mentioned before will be selected and created. The prepared question pool will be presented to the expert opinion of 11 people and the scale questions will be clarified. The pilot study of the scale will be conducted with a total of 40 patients, 10 participants for each patient group. After the pilot study, item analyses and exploratory factor analysis (EFA) analysis will be performed with a sample size of 5 times the number of questions in the item pool with acute and chronic pain patients. Afterwards, confirmatory factor analysis (CFA) analysis will be performed for the factor structure obtained with a sample size 10 times the number of remaining items (a second study). In addition, a correlation analysis study will be performed with the new scale and TSK scale for test-retest reliability (ICC) and validity. , Inclusion criteria: Young, middle-aged, neurologic, geriatric patients aged 18-70 years with chronic musculoskeletal pain problems after acute injury or surgery will be included.

Exclusion criteria: illiterate patients, patients with cognitive and cooperation problems will not be included in the study.

When the new scale development process is completed, validation studies of the scale on neurological and geriatric patient population will continue. The project outputs are planned to be published as scientific articles within the scope of SCI and as papers in international and national congresses. The project article will be translated into other languages abroad and cultural adaptations will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Young, middle-aged, neurologic, geriatric patients
* aged 18-70 years with chronic musculoskeletal pain problems after acute injury or surgery will be included.

Exclusion Criteria:

* patients with cognitive and cooperation problems will not be included in the study.
* illiterate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of male and female patients aged 18-70 years with complaints of acute and chronic pain due to musculoskeletal problems.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
The pilot study of the scale will be conducted with a total of 40 patients, 10 participants for each patient group. | Up to one month
item analyses and exploratory factor analysis (EFA) analysis will be performed with a sample size of 5 times the number of questions in the item pool with acute and chronic pain patients. | Up to one month

CONTACTS AND LOCATIONS:
Overall Officials: Ayhan Parmaksız, PhD, Principal Investigator — İstanbul Sağlık ve Teknoloji Üniversitesi
Locations (1):
- Atılım University, Ankara, Turkey (Türkiye)